CLINICAL TRIAL: NCT00586703
Title: Safety Trial of Natural Killer (NK) Cell Donor Lymphocyte Infusions (DLI) From 3-5/6 Human Leukocyte Antigen (HLA) Matched Family Member Following Nonmyeloablative Allogeneic Stem Cell Transplantation (ASCT)
Brief Title: Safety Trial of NK Cell DLI 3-5/6 Family Member Following Nonmyeloablative ASCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005123
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma
Keywords: Stem cell transplant; mismatched donor; NK infusion
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NK-CD56 (Experimental): NK Cell infusion using CD56 monoclonal antibody following nonmyeloablative SCT from mismatched donors
  Interventions: Device: NK-CD56

INTERVENTIONS:
Device: NK-CD56 — NK Cell infusion using CD56 monoclonal antibody following nonmyeloablative SCT from mismatched donors: The cells from leukapheresis will be NK selected using a CD56 antibody and a cell column system provided by Miltenyi Biotec. The target cell dose for each NK cell infusion will be up to 1 X 10(7) CD56+ cells/kg patient weight with less than 0.5 X 10(6) CD3+ cells/kg patient weight. The first NK cell infusion will be administered 6 weeks post transplant in patients who have ≤ grade II aGVHD at the time of infusion. Patients will be evaluated for toxicity and response until 20 weeks after the last NK Infusion.

SUMMARY:
Evaluate the safety of natural killer (NK) cell infusion using CD56 monoclonal antibody selected with Miltenyi Biotec system following nonmyeloablative stem cell transplantation (SCT) from mismatched donors. This pilot study will evaluate toxicity including mortality, occurrence of acute graft versus host disease (aGVHD) and other severe toxicity.

DETAILED DESCRIPTION:
The use of non-selected donor lymphocyte infusions (DLIs) (to help early immune recovery and induce antitumor response) following nonmyeloablative allogeneic stem cell transplantation (ASCT) is also complicated by the risk of acute graft versus host disease (aGVHD) with 30-40% of patients experiencing grade III-IV aGVHD. Data suggests that the use of natural killer (NK) cells (instead of nonselected DLIs) in this setting may mediate a graft versus tumor (GVT) effect independently of aGVHD.

This pilot study is designed to evaluate the efficacy and toxicity of donor natural killer (NK) cell selection and infusion following nonmyeloablative allogeneic stem cell transplantation from mismatched donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with who have undergone a non-myeloablative allogeneic transplant, using a 3-5/6 HLA matched sibling donor. Measureable disease is not needed at study entry.
* Performance status must be Karnofsky 50-100%.
* Donor cellular engraftment of at least 2.5% from the non-myeloablative procedure.
* ≤ Grade 2 acute GVHD at time of infusion of NK cell infusion. Patients with treated acute GVHD must be on a stable dose of therapy (no increase in immunosuppressive therapy for the 2 weeks before planned NKI). The dosage/level of immunosuppressive therapy at the time of NKI should be no greater than 1 mg/kg of prednisone daily or mycophenolate 1000 mg bid daily or cyclosporine with a target level of 200 or equivalent.
* Estimated survival at least 8 weeks.
* Age > or equal to 18 years of age.

Exclusion Criteria:

* Pregnant or lactating women,
* Patients with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise tolerance to this protocol.
* Patients who had biopsy proven overall Grade 4 GVHD lasting longer than 7 days, from the non-myeloablative therapy, are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-04; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke University Health Systems
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

REFERENCES:
- [Result] Rizzieri DA, Storms R, Chen DF, Long G, Yang Y, Nikcevich DA, Gasparetto C, Horwitz M, Chute J, Sullivan K, Hennig T, Misra D, Apple C, Baker M, Morris A, Green PG, Hasselblad V, Chao NJ. Natural killer cell-enriched donor lymphocyte infusions from A 3-6/6 HLA matched family member following nonmyeloablative allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2010 Aug;16(8):1107-14. doi: 10.1016/j.bbmt.2010.02.018. Epub 2010 Feb 24. PMID 20188202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 Patients were recruited through the Adult Bone Marrow Transplant Program at Duke University Medical Center. Recruitment began in April, 2005 and ended in March, 2011. Patients who met the eligibility criteria were approached about the study and informed consent was conducted for those who agreed.
Pre-assignment Details: Prior to donor lymphocyte infusion (DLI), disease state was documented:
  Complete history Physical exam Performance status Routine lab tests Radiographic tests Subjects didn't continue with treatment with disease progression. 2 subjects withdrew consent; 1 had graft versus host disease; 1 died; 1 subject's donor didn't yield enough cells.
Groups:
- Experimental: NK-CD56: NK Cell infusion using CD56 monoclonal antibody following nonmyeloablative SCT from mismatched donors
  NK Cell Infusion following SCT from mismatched donors : The cells from leukapheresis will be NK selected using a CD56 antibody and a cell column system provided by Miltenyi Biotec. The target cell dose for each NK cell infusion will be up to 1 X 10(7) CD56+ cells/kg patient weight with less than 0.5 X 10(6) CD3+ cells/kg patient weight. The first NK cell infusion will be administered 6 weeks post transplant in patients who have ≤ grade II aGVHD at the time of infusion. Patients will be evaluated for toxicity and response until 20 weeks after the last NK Infusion.
Period: Overall Study
Arm/Group | Experimental: NK-CD56
Started | 16
Completed | 4
Not Completed | 12
Not completed — Death | 12

BASELINE CHARACTERISTICS:
Population: Participants who were eligible for study.
Groups:
- Experimental: NK-CD56: Natural Killer (NK) Cell infusion using CD56 monoclonal antibody following nonmyeloablative stem cell transplant (SCT) from mismatched donors
  NK Cell Infusion following SCT from mismatched donors: The cells from leukapheresis will be NK selected using a CD56 antibody and a cell column system provided by Miltenyi Biotec. The target cell dose for each NK cell infusion will be up to 1 X 10(7) CD56+ cells/kg patient weight with less than 0.5 X 10(6) CD3+ cells/kg patient weight. The first NK cell infusion will be administered 6 weeks post transplant in patients who have ≤ grade II acute graft-versus host disease (aGVHD) at the time of infusion. Patients will be evaluated for toxicity and response until 20 weeks after the last NK Infusion.
Arm/Group | Experimental: NK-CD56
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Evaluate the safety of NK cell infusion using CD56 monoclonal antibody following nonmyeloablative stem cell transplantation from mismatched donors: Toxicity including mortality, occurrence of acute graft versus host disease (aGVHD) and other severe toxicity.
Time Frame: 8 weeks
Population: Participants who were able to receive infusion.
Measure: Number; unit: participants
Arm/Group | Experimental: NK-CD56
Number analyzed (Participants) | 16
participants
  Acute Graft versus Host Disease (aGvHD) | 8
  Post-transplant lymphoproliferative disorder | 2

2. Secondary Outcome: Efficacy - Overall Survival
Description: Evaluate the efficacy of the regimen in terms of overall survival (OS).
Time Frame: 7 years
Population: Participants who completed infusion.
Measure: Mean (Full Range); unit: months
Arm/Group | Experimental: NK-CD56
Number analyzed (Participants) | 16
months | 27 [4 to 84]

ADVERSE EVENTS:
Time Frame: Patients shall be monitored for toxicity and Graft versus Host Disease every other week until 8 weeks after the last Natural Killer cell Infusion and after that, every 4 weeks for 12 more weeks.
Arm/Group | Experimental: NK-CD56
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: NK-CD56 (N=16)
Failure to Engraft (Investigations) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Supraventricular and nodal arrhythmia
Atrial Flutter (Cardiac disorders) | 1 (1) — Supraventricular and nodal arrhythmia
Dermatology - Skin (other) (Skin and subcutaneous tissue disorders) | 1 (1) — Squamous cell carcinoma - left chest
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — desquamation - contact dermatitis on neck and face
Diarrhea (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1) — ulcerative esophagitis
Hemorrhagic Cystitis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage - GU (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (2) — fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C
Infection - other (Infections and infestations) | 1 (1) — Cytomegalovirus Retinitis
Infection-bacterial with grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 5 (6) — C-diff; Gram-rod bacteria; Methicillin-resistant Staphylococcus aureus (MRSA); Klebsiella; E-coli; Bacillus and Coag Negative Staph
Infection-bacterial with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 3 (5) — Osteomyelitis; Pseudomonas bacteremia; Staph; Enterococcus
Infection-viral without febrile neutropenia (Infections and infestations) | 3 (3) — Cytomegalovirus; Viremia; Parainfluenza
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
AST; SGOT (Metabolism and nutrition disorders) | 1 (1) — Aspartate transaminase; serum glutamic oxaloacetic transaminase
Creatinine (Metabolism and nutrition disorders) | 1 (1) — 4.3 mg/dl
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1) — Motor neuropathy
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Post-transplant lymphoproliferative disorder
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Blood/Bone Marrow - Blast Crisis (Blood and lymphatic system disorders) | 1 (1) — Relapsed Acute myeloid leukemia
Infection-viral with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 5 (7) — Cytomegalovirus; Viremia; Polyoma; Herpes; Varicella Zoster
Infection-viral with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 7 (11) — Adenovirus; Cytomegalovirus; Parainfluenza; Polyoma; Human Herpes Virus 6; Viremia
Hypervolemia (Blood and lymphatic system disorders) | 1 (1)
Infection-bacterial without febrile neutropenia (Infections and infestations) | 1 (1) — Gram positive Cocci bacteria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes